CLINICAL TRIAL: NCT00268866
Title: Danish Quality Assurance Project on Diagnosis and Treatment of COPD in Outpatient Lung Clinics
Brief Title: Danish Quality Assurance Project on Diagnosis and Treatment of Chronic Obstructive Pulmonary Disease (COPD) in Outpatient Lung Clinics
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Other Study IDs: 205.367
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

INTERVENTIONS:
Behavioral: Education

SUMMARY:
Danish Quality Assurance Project on Diagnosis and Treatment of COPD in Outpatient Lung Clinics

DETAILED DESCRIPTION:
Study Hypothesis:

Comparison(s):

none

ELIGIBILITY:
Inclusion Criteria:

* Outpatient with the diagnosis or referral diagnosis of COPD.
* COPD must be the primary reason for this outpatient contact (for both new patients and controls).

Exclusion Criteria:

* Any co-morbidity that hampers the diagnosis and treatment of COPD in accordance with the COPD guidelines used locally (e.g. malignant disease, dementia or sequelae of apoplexy).
* Asthma without the presence of COPD

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1820
Dates: Study Completion 2007-01

PRIMARY OUTCOMES:
To optimise the diagnosis and treatment of COPD via a quality assurance project
Increase the knowledge and use of diagnostic tools and treatment options
Increase focus on COPD comorbidity

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Denmark A/S